CLINICAL TRIAL: NCT03264313
Title: A Prospective, Placebo-controlled, Randomized, Double-blind Study to Evaluate the Safety and Efficacy of the Use of Deep Transcranial Magnetic Stimulation (dTMS) on Smoking Cessation.
Brief Title: Deep Transcranial Magnetic Stimulation (dTMS) to Induce Smoking Cessation
Acronym: SmokCessdTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Manoel Jacobsen Teixeira, Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35068014400000068
Record Dates: First submitted 2017-08-16; First posted 2017-08-29 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Smoking Cessation; Transcranial Magnetic Stimulation
Keywords: tobacco; Smoking Cessation; TMS; Neuromodulation; transcranial magnetic stimulation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- dTMS active (Active Comparator): patients undergoing of dTMS real
  Interventions: Device: Deep Transcranial Magnetic Stimulation
- dTMS Sham (Sham Comparator): patients undergoing to placebo dTMS
  Interventions: Device: Deep Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation — Patients undergoing of Deep Transcranial Magnetic Mtimulation (dTMS) for smoking cessation
  Other Names: dTMS

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of dTMS used as a tool for the smoking cessation; therefore, the subjects will be randomized to be treated on the active group or to receive placebo stimulation.

DETAILED DESCRIPTION:
Smoking is the leading cause of preventable deaths in the world. Tobacco use causes more than 5 million deaths per year worldwide.

Among interventions methods that have been found to be effective, the medications are the most promising, using drugs such as Varenicline and Bupropion. Nicotine replacement therapy (NRT) shows results in combination to these drugs.

Alternative approaches to smoking cessation such as acupuncture, hypnosis, smokeless tobacco, electronic cigarettes are not legitimated smoking cessation tools; given that scientific studies showed no difference between these methods and placebo, or yet no rigorous peer-reviewed studies have been conducted.

On the neuromodulation field, Repetitive Transcranial Magnetic Stimulation (rTMS) appears as a new possibility to treat this serious condition.

The rTMS is a non-invasive method of stimulating cortical neurons. Repetitive TMS has been tested as a treatment of various neuropsychiatric disorders associated with cortical excitability disfunctions.

Several lines of evidence suggest that rTMS over the prefrontal cortex (PFC) can affect processes involved in nicotine addiction. First, animal studies demonstrated that rTMS to the frontal regions of rats enhanced release of dopamine in the hippocampus and NAc . Moreover, high-frequency rTMS of the human prefrontal cortex (PFC) has been shown to induce dopamine release in the caudate nucleus. Hence, it has been suggested that high-frequency rTMS may be useful in disorders associated with subcortical dopamine dysfunction, such as addiction.

Several human studies have begun to evaluate the effects of rTMS protocols applied to the PFC on drug craving and consumption in nicotine. Johann and colleagues reported decreased levels of tobacco craving after single rTMS session over the left dorsolateral prefrontal cortex (DLPFC). In addition, a single session of rTMS over the right DLPFC can reduce cocaine craving. Eichhammer and colleagues in a cross-over, double-blind, placebo-controlled study demonstrated a reduction in cigarette consumption (measured 6 hours following the treatment) but craving levels remained unchanged after two rTMS sessions over the left DLPFC. Amiaz and collegues found that 10 days of high-frequency rTMS over the DLPFC reduced cigarette consumption and nicotine dependence. In addition, the rTMS blocked craving induced by smoking cues. However, the effect tended to dissipate after the 10 daily sessions and the reduction in cigarette consumption was not significant 6 months after treatment termination. Moreover, only 10% among those who responded to the treatment had totally quit smoking. Li et al treated subjects with real high-frequency rTMS or sham TMS over the DLPFC in two visits with 1 week between visits. The participants received cue exposure before and after rTMS. Stimulation of the left DLFPC with real rTMS reduced craving significantly from baseline. When compared with neutral cue craving, the effect of real TMS on cue craving was significantly greater than the effect of sham TMS. Rudction in subjective craving induced by TMS correlated positively with higher Fagerström Test for Nicotine Dependence score and more cigarettes smoked per day. These four studies demonstrate that high-frequency rTMS of the DLPFC can attenuate nicotine consumption and craving. However, the significance and duration of these effects are limited and further investigation is required to identify the appropriate stimulation parameters and targets needed to enhance the effectiveness of such treatment.

One possible reason for these partial effects on nicotine consumption might be the superficial magnetic stimulation induced by the figure-8 coil, which does not reach into the deep layers of the cortex. It is known that nicotine addiction involves various areas of the brain reward system. Most of them are deeper than the superficial layers of the cortex, like the anterior cingulated, orbitofrontal cortex, nucleus accumbens, and amygdala.

Another area of interest which was not stimulated using the superficial rTMS is the insula. A recent study explored the role of insula damage in addiction. In a retrospective design, assessing changes in cigarette smoking after brain damage, results revealed that smokers with brain damage involving the insula were significantly more likely to undergo a disruption of smoking addiction than smokers with brain damage not involving the insula. This finding is consistent with the crucial role of the insula in cravings for food, cocaine and cigarettes, as reported by neuroimaging studies, and with the role of the insula in processes related to decision-making. Therefore stimulating the insula and the deeper layers of the lateral PFC could be substantially more effective in treating nicotine addiction.

Deep Transcranial Magnetic Stimulation (dTMS) is a new form of rTMS which allows direct stimulation of deeper neuronal pathways than standard rTMS using the Brainsway's new H-coils. In this study we will apply the dTMS using the H-ADD, which is designed to reach deeper brain areas related to the control of motivation, reward and pleasure, specifically, fibers connecting the DLPFC and the insula.

Given these theoretical, animal and preliminary human data, we hypothesized that a course of deep high-frequency, using a specific coil for deep stimulation (H-ADD) over the right and left lateral PFC and insula, may reduce impulsivity, nicotine dependence and craving for cigarettes in response to smoking-related cues.

ELIGIBILITY:
Inclusion Criteria:

* Current heavy (> 10 cigarettes / day) and chronic smokers (who have smoked for more than 1 year, with no abstinence greater than 3 months during the past year);
* Motivated to quit smoking;
* Capable to receive TMS treatment (satisfactory answers at the Safety Questionnaire for Transcranial Magnetic Stimulation);
* Consent report signed by the study participant.

Exclusion Criteria:

* Using nicotine replacement therapy or drugs to aid in smoking cessation (eg Bup, etc.) or dealing with behavioral therapy for smoking cessation.
* Functional or cognitive disorder, diagnosis according to DSM-5.
* Psychiatric Disorder active in the last year, according to DSM-5 (Axis I). Exception to depressive and anxious disorders, provided that in a stable condition.
* Substance or drug abuse or dependency in the current or in the last year prior to selection.
* Subjects who smoke any other type of tobacco or substances.
* Subjects with a high risk of violence or suicide assessed during the interview.
* Subjects suffering from any physical instability such as high blood pressure (> 150 mmHg systolic / diastolic> 110 mmHg) or acute or unstable heart disease.
* History of epilepsy or seizure (EXCEPT those therapeutically induced by ECT).
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head injury or trauma with loss of consciousness for > 5 minutes.
* History of any metal in the head (outside the mouth).
* Metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* Individuals with a significant neurological disorder or insult;
* Subjects suffering from frequent and severe migraine headaches.
* Subjects suffering from significant hearing loss.
* Subjects taking pro-convulsant medications (e.g., antipsychotic medications).
* Previous treatment with TMS.
* Subjects who cannot communicate reliably with the investigator or who are not likely to cope with the requirements of the experiment.
* Participation in a clinical trial within the last 30 days before the beginning of this clinical trial or similar participation in another clinical trial.
* Known or suspected pregnancy or lactation.
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Decrease on Monoximetry level | before each session at phase 1 (6 weeks = sessions from 1 to 18)
  The researchers will perform the measurement of the rate of expired carbon monoxide through a monoximeter.

SECONDARY OUTCOMES:
Changes on Cotinine blood level | at session 1 and after session 18 (6 weeks)
  The test uses a device that measures the levels of cotinine through a drop of blood obtained from a slight bite on the tip of the participant's finger.

OTHER OUTCOMES:
Diary | once a week at the first phase: 6 weeks
  Self reported daily number of cigarettes

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Marcolin, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Incor - Instituto do Coração do HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scholz JR, Bellini BB, Ziotti SDV, Abe TO, Arnaut D, Alberto RL, Marcolin MA, Tonstad S. Cue-Restricted Smoking as a behavioral adjunct for smoking cessation: Observational sub-analysis of a randomized trial of deep transcranial magnetic stimulation. Tob Prev Cessat. 2025 Oct 3;11. doi: 10.18332/tpc/209189. eCollection 2025. PMID 41048875